CLINICAL TRIAL: NCT06649578
Title: Comparing Bariatric Surgery Outcomes in Predominantly High-Risk Asian Patients to Global Benchmarks: Insights From a Decade-Long Cohort Study of 1016 Patients
Brief Title: Comparing Bariatric Surgery Outcomes in Predominantly High-Risk Asian Patients to Global Benchmarks
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022/00303
Record Dates: First submitted 2024-10-08; First posted 2024-10-21 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2023-07

CONDITIONS: Bariatric Surgery; Cost of Care; Complications
Keywords: Metabolic-bariatric surgery; Costs; Outcomes; Comprehensive Complication Index; Asians
MeSH Terms: interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metabolic-Bariatric Surgery: Patients undergoing Metabolic-Bariatric Surgery are divided into either Laparoscopic Sleeve Gastrectomy (LSG), Roux-en-Y Gastric Bypass (RYGB) or One-Anastomosis Gastric Bypass (OAGB).
  Interventions: Procedure: Metabolic-bariatric surgery

INTERVENTIONS:
Procedure: Metabolic-bariatric surgery — Our study is conducted in a predominantly high-risk Asian population that will be undergoing metabolic-bariatric surgery. The types of surgery can be divided into Laparoscopic Sleeve Gastrectomy (LSG), Roux-en-Y Gastric Bypass (RYGB) or One-Anastomosis Gastric Bypass (OAGB).

SUMMARY:
While metabolic-bariatric surgery is a safe and well-established surgery, complications do occur and can have significant impact on the patient. With the study, the investigators aim to establish the proportion of patients that will have complications and understand what the impact of complications are on costs.

DETAILED DESCRIPTION:
Complications after metabolic-bariatric surgery can be catastrophic and have significant impact on costs, morbidity, and mortality. As current global benchmarks for complications rates in MBS are based on standard risk patients in western populations, the benchmark complication rates in high-risk patients and Asian populations are unknown. The investigators aim to evaluate the incidence of complications in 1016 consecutive patients and the impact of complications on costs.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were patients who underwent either primary or revisional MBS comprising Laparoscopic Sleeve Gastrectomy (LSG), Roux-en-Y Gastric Bypass (RYGB) or One-Anastomosis Gastric Bypass (OAGB).

Exclusion Criteria:

* Patients under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our patients are consecutive patients that underwent metabolic-bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1016 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Anastomotic Leak | From completion of surgery till post-operative 90 days
  90 Day Post-Operative Complications
Number of Participants with Bleeding | From completion of surgery till post-operative 90 days
  90 Day Post-Operative Complications
Number of Participants with Perforation | Time Frame: From completion of surgery till post-operative 90 days
  90 Day Post-Operative Complications
Number of Participants with Collection | Time Frame: From completion of surgery till post-operative 90 days
  Collection includes hematoma, pus, serous fluids. Outcome measured to 90 Day Post-Operative.
Number of Participants with Hospital Readmission | From completion of surgery till post-operative 90 days
  Any readmission to hospital from completion of surgery till post-operative 90 days
Number of Participants with Reoperation | From completion of surgery till post-operative 90 days
  Any reoperation due to any complications from completion of surgery till post-operative 90 days

SECONDARY OUTCOMES:
Total Costs of Bariatric Surgery (USD) | From completion of surgery till post-operative 90 days
  Total costs of all events that occur from surgery till post-operative 90 days will be included. Costs will be extracted from hospital records.
Time to surgical intervention (hr) | From completion of surgery till 90 days post-operative
  Time to surgical intervention for patients requiring surgical treatment for post-operative complications. Time will be extracted from surgical records
Number of Participants with Total Parental Nutrition Requirement | From completion of surgery till post-operative 90 days
  Use of Total Parental Nutrition during 90 Day Post-Operative
Number of Participants with Blood Transfusion | From completion of surgery till post-operative 90 days
  Any blood transfusion given from completion of surgery till post-operative 90 days
Length of Stay (Days) | From completion of surgery till hospital discharge assessed up to post-operative 90 days
  Length of hospital stay from index operation to hospital discharge
Number of Participants with Emergency Department Attendance | From completion of surgery till post-operative 90 days
  Any Emergency Department Attendance from completion of surgery till post-operative 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Asim Shabbir, MBBS, FRCS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon reasonable request towards corresponding author.

REFERENCES:
- [Result] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Result] Gero D, Raptis DA, Vleeschouwers W, van Veldhuisen SL, Martin AS, Xiao Y, Galvao M, Giorgi M, Benois M, Espinoza F, Hollyman M, Lloyd A, Hosa H, Schmidt H, Garcia-Galocha JL, van de Vrande S, Chiappetta S, Menzo EL, Aboud CM, Luthy SG, Orchard P, Rothe S, Prager G, Pournaras DJ, Cohen R, Rosenthal R, Weiner R, Himpens J, Torres A, Higa K, Welbourn R, Berry M, Boza C, Iannelli A, Vithiananthan S, Ramos A, Olbers T, Sepulveda M, Hazebroek EJ, Dillemans B, Staiger RD, Puhan MA, Peterli R, Bueter M. Defining Global Benchmarks in Bariatric Surgery: A Retrospective Multicenter Analysis of Minimally Invasive Roux-en-Y Gastric Bypass and Sleeve Gastrectomy. Ann Surg. 2019 Nov;270(5):859-867. doi: 10.1097/SLA.0000000000003512. PMID 31592894